CLINICAL TRIAL: NCT04918901
Title: Comparative Analysis of Clinical Indicators and Imaging Changes of Severe COVID-19
Brief Title: Comparative Analysis of Clinical Parameters and Radiographic Changes of Severe COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: xp2020-355
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Severe COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe COVID-19: Comparative Analysis of Clinical Parameters and Radiographic Changes
  Interventions: Combination Product: NO Severe COVID-19

INTERVENTIONS:
Combination Product: NO Severe COVID-19 — Non-severe and critically ill patients with COVID-19

SUMMARY:
Novel Coronavirus Pneumonia (COVID-19) is the pneumonia caused by the 2019 novel coronavirus infection. Critically ill patients with this disease develop dyspnea and hypoxemia, and even further aggravate acute respiratory distress syndrome, septic shock, coagulation dysfunction, and multiple organ failure. Since February 15, 2020, the 171-member medical team of the Second Affiliated Hospital of Zhejiang University School of Medicine has taken over the Intensive Care Unit of the Cancer Center of the Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology and the Intensive Care Unit of the West Hospital of Union Hospital to carry out severe and critical care. Treatment of patients with new coronary pneumonia. In clinical practice, combined with the changes in chest CT imaging of severe COVID-19 patients, it has been found that some laboratory indicators of severe patients can effectively judge the clinical prognosis and outcome of patients, but there is no relevant retrospective study with large sample size so far.

DETAILED DESCRIPTION:
Novel Coronavirus Pneumonia (COVID-19) is the pneumonia caused by the 2019 novel coronavirus infection. Critically ill patients with this disease develop dyspnea and hypoxemia, and even further aggravate acute respiratory distress syndrome, septic shock, coagulation dysfunction, and multiple organ failure. Since February 15, 2020, the 171-member medical team of the Second Affiliated Hospital of Zhejiang University School of Medicine has taken over the Intensive Care Unit of the Cancer Center of the Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology and the Intensive Care Unit of the West Hospital of Union Hospital to carry out severe and critical care. Treatment of patients with new coronary pneumonia. In clinical practice, combined with the changes in chest CT imaging of severe COVID-19 patients, it has been found that some laboratory indicators of severe patients can effectively judge the clinical prognosis and outcome of patients, but there is no relevant retrospective study with large sample size so far.

In April 16, 2020, the investigators submitted the research project, comparative analysis of clinical parameters and radiographic changes of severe COVID-19, to human subject research ethics committee of Second Affiliated Hospital, School of Medicine, Zhejiang University. The research process began after the committee for approval in May 2020.

In this study, by comparing the changes in chest CT imaging of patients with severe COVID-19, the investigators analyzed the effects of some clinical indicators on the prognosis and outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19 patients who meet the criteria for confirmed cases in the "New Coronavirus Pneumonia Diagnosis and Treatment Plan (Trial Seventh Edition)";
2. The clinical classification is severe and critical.

Exclusion Criteria:

1. Patients who died within 72 hours of admission;
2. Patients who cannot be transferred to chest CT imaging due to their medical conditions.

Ages: 34 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe and critical COVID-19 patients admitted to the Intensive Care Unit of the Cancer Center of Union Hospital of Tongji Medical College of Huazhong University of Science and Technology and the Intensive Care Unit of West Hospital of Union Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Lactic acid measurement in the blood gas results indirectly reflects the body's respiratory function, and it can also reflect the degree of metabolic acidosis in the body. | up to 6 weeks
  Weekly monitoring of blood gas analysis in severe COVID-19 patients. Lactic acid measurement in the blood gas results indirectly reflects the body's respiratory function, and it can also reflect the degree of metabolic acidosis in the body.
The possibility of inflammatory response in patients with large lymphocytes COVID-19 levels were significantly reduced. | up to 6 weeks
  Weekly monitoring of blood routine in severe COVID-19 patients. The possibility of inflammatory response in patients with large lymphocytes COVID-19 levels were significantly reduced.
C-reactive protein（CRP） rises rapidly, but the rise is moderate, which can be used as an auxiliary diagnostic index for sepsis after COVID-19. | up to 6 weeks
  Weekly monitoring of C-reactive protein （CRP）in severe COVID-19 patients. After the new coronavirus infection, CRP rises rapidly, but the increase is moderate, which is an auxiliary diagnostic index for sepsis.
Procalcitonin（PCT) is a diagnostic indicator of bacterial sepsis after COVID-19. | up to 6 weeks
  Weekly monitoring of procalcitonin in severe COVID-19 patients. After the new coronavirus infection, PCT has high specificity, but the level does not increase or slightly increases, which is a diagnostic indicator of bacterial sepsis.
The continuous decline of cluster of differentiation 4+ T cells(CD4+) and cluster of differentiation 8+ T cells (CD8+ ) should be alert to the deterioration of COVID-19. | up to 6 weeks
  Weekly monitoring of CD4+/CD8+ in severe COVID-19 patients. The continuous decline of CD4+ and CD8+ T cells should be alert to the deterioration of the disease.
The progressive rise of interleukin-6 (IL-6) as a clinical warning indicator for the deterioration of COVID-19. | up to 6 weeks
  Weekly monitoring of interleukin-6 in severe COVID-19 patients. The level of IL-6 increase is consistent with the severity of the disease. Once the disease is under control, it will drop rapidly; if it does not decrease rapidly after treatment, it often indicates a poor prognosis. The notification of the diagnosis and treatment plan for severe and critical cases of new coronavirus pneumonia (the second version on trial) has clearly identified the progressive rise of IL-6 as a clinical warning indicator for the deterioration of the disease.
Chest computer tomography (CT) can reflect the progress of the disease, and may have a certain prompting effect on the prognosis of COVID-19 patients. | up to 6 weeks
  Weekly monitoring of chest CT imaging of patients with severe COVID-19. COVID-19 is highly contagious, chest CT manifestations are diverse, with multiple ground glass shadows in both lungs with or without partial solidification as the main feature, mainly subpleural distribution, as the course of the disease progresses, CT manifestations gradually increase with the time of onset. At the same time, CT semi-quantitative scores can reflect the progress of the disease, and may have a certain prompting effect on the prognosis of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, Professor, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Neuroscience care unit, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided